CLINICAL TRIAL: NCT03525574
Title: A Phase 3, Open-label Study Evaluating the Long-term Safety and Efficacy of VX-445 Combination Therapy in Subjects With Cystic Fibrosis Who Are Homozygous or Heterozygous for the F508del Mutation
Brief Title: A Study Evaluating the Long-term Safety and Efficacy of VX-445 Combination Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX17-445-105; 2018-000185-11 (EudraCT Number)
Expanded Access: NCT04058210 (Approved for marketing)
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX/TEZ/IVA (Experimental): Treatment Period: Participants received ELX 200 milligram (mg) once daily (qd)/TEZ 100 mg qd/IVA 150 mg every 12 hrs (q12h) in the treatment period for 192 weeks.
  Extension Period: Participants from certain countries participated in extension period and continued to receive ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the extension period for 48 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination (FDC) tablet for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
The study evaluates the long-term safety and tolerability of VX-445 in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are homozygous or heterozygous for the F508del mutation

ELIGIBILITY:
Inclusion Criteria:

* Completed study drug treatment in a parent study i.e.VX17-445-102 (NCT03525444) and VX17-445-103 (NCT03525548); or had study drug interruption(s) in a parent study but completed study visits up to the last scheduled visit of the Treatment Period in the parent study.

Exclusion Criteria:

* History of drug intolerance in a parent study that would pose an additional risk to the subject in the opinion of the investigator.
* Current participation in an investigational drug trial (other than a parent study)

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (52):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Miller Children's Hospital / Long Beach Memorial, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Gateway Medical Center, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Florida, Shands Hospital, Gainesville, Florida
  - Joe DiMaggio Cystic Fibrosis & Pulmonary Center, Hollywood, Florida
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Tampa General Hospital Cardiac and Lung Transplant Clinic, Tampa, Florida
  - Children's Specialty Services at North Druid Hills, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Cystic Fibrosis Center, Children's Hospital of Illinois at OSF Saint Francis Medical Center, Peoria, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - Maine Medical Partners, Portland, Maine
  - Massachusetts General Hospital Cystic Fibrosis Center Clinical Research Center, Boston, Massachusetts
  - Harper University Hospital, Detroit, Michigan
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Billings Clinic Hospital, Billings, Montana
  - Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - UNM Clinical and Translational Science Center, Albuquerque, New Mexico
  - The Cystic Fibrosis Center, Mount Sinai Beth Israel, New York, New York
  - New York Medical College, Valhalla, New York
  - UNC Marsico Clinical Research Center, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - UC Health Holmes, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Toledo Children's Hospital/Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Vermont Lung Center, Colchester, Vermont
  - University of Virginia Primary Care Center, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital of Richmond at VCU, Children's Pavilion, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - CTSI Adult Translational Research Unit/Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Australia (5):
  - Women & Children's Hospital, North Adelaide
  - The Royal Children's Hospital, Parkville
  - Mater Misericordiae Ltd, South Brisbane
  - The Children's Hospital at Westmead, Westmead
  - Westmead Hospital, Westmead
- Austria (4):
  - University of Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medizinische Universitat Wien, Vienna
- Belgium (5):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (6):
  - University of Calgary Medical Clinic of the Foothills Medical Centre, Calgary
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - Centre Hospitalier De L'Universite Laval, Québec
  - The Hospital for Sick Children, Toronto
  - British Columbia's Children's Hospital, Vancouver
  - St. Paul's Hospital, Vancouver
- Czechia (2):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni nemocnice v Motole, Prague
- France (7):
  - Centre Hospitalier Lyon Sud, Benite Cedex
  - Groupe Hospitaler Pellegrin, CHU De Bordeaux, Bordeaux
  - CHU Marseille - Hopital Nord, Marseille
  - CHU de Nice - Hopital Pasteur, Nice
  - Hopital Cochin, Paris
  - CHU de Rouen - Hopital Charles Nicolle, Rouen
  - Hopital Foch (Suresnes), Hopital Foch, Adultes, Suresnes
- Germany (7):
  - Friedrich-Alexander University of Erlangen-Nuremberg, University Children's Hospital, Erlangen
  - Justus-Leibig-Universitat Zentrum fur Kinderheilkunde und Jugendmedizin, Giessen
  - Hannover Medical School, Hanover
  - Johannes Gutenberg-Universitaet, Mainz
  - Dr. von Haunersches Kinderspital, München
  - Universitaetsklinikum Tuebingen Klinik fuer Kinder- und Jugendmedizin, Tübingen
  - University Hospital Wuerzburg, Würzburg
- General Hospital of Attika "Sismanoglio"(Adult CF center, NHS), Marousi, Greece
- Italy (7):
  - Azienda Ospedaliero Universitaria Ospendali Riuniti, Ancona
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico, Genova
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Centro Regionale Fibrosi Cistica, A.O. Ospedale San Carlo, Potenza
  - Azienda Ospedaliera di Verona-Ospedale Civile Maggiore, Verona
- Netherlands (5):
  - Academic Medical Center, Amsterdam
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Heidelberglaan
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague
- Karolinska Universitetssjukhuset, Huddinge, Stockholm, Sweden
- United Kingdom (8):
  - Belfast City Hospital, Belfast
  - Heart of England NHS Foundation Trust, Birmingham Heartlands Hospital, Birmingham
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter NHS Foundation Trust, Royal Devon and Exeter Hospital, Exeter
  - Leeds General Infirmary, Leeds
  - King's College Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Daines CL, Polineni D, Tullis E, Costa S, Linnemann RW, Mall MA, McKone EF, Quon BS, Ringshausen FC, Selvadurai H, Taylor-Cousar JL, Withers NJ, Sawicki GS, Lee T, Ahluwalia N, Morlando Geiger J, Jennings M, Tan YV, Waltz D, Ramsey B, Griese M; VX17-445-105 Study Group. Long-Term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor in Adults and Adolescents with Cystic Fibrosis and at Least One F508del Allele: A Phase 3 Open-Label Extension Study. Am J Respir Crit Care Med. 2025 Oct;211(10):1901-1914. doi: 10.1164/rccm.202411-2231OC. PMID 40209082
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted as a single period i.e. treatment period in countries including United States (US) with commercially-available ELX/TEZ/IVA. The regional protocol for other countries without commercially-available ELX/TEZ/IVA was amended so that participants in these countries had the opportunity to participate for up to an additional 48 weeks in extension period.
Pre-assignment Details: A total 507 participants were enrolled in this study from the parent studies VX17-445-102 (NCT03525444) and VX17-445-103 (NCT03525548). One participant was enrolled but did not receive any dose in this study.
Groups:
- Additional Participants for Cumulative TC Efficacy Set: This reporting arm represents the three additional participants in Cumulative TC Efficacy Set 102/105 from parent study 102 which were not not enrolled in this study, but were included in the Cumulative TC efficacy 102/105 analysis set.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA | Additional Participants for Cumulative TC Efficacy Set
Started | 507 | 3
Open-Label Safety Set (OL-SS) | 506 (The Open-Label Safety Set (OL-SS) included all participants who had received at least 1 dose of study drug in this open label study.) | 0
OL-FAS 102/105 | 399 (The OL Full Analysis Set (FAS) 102/105 included participants enrolled from parent study 102 who received at least 1 dose of study drug in this open label study.) | 0
OL-FAS 103/105 | 107 (The OL-FAS 103/105 included participants enrolled from parent study 103 who received at least 1 dose of study drug in this open label study.) | 0
Cumulative Triple Combination (TC) Efficacy Set 102/105 | 400 (Cumulative TC Efficacy Set 102/105 included all participants who were randomized to TC ELX/TEZ/IVA and received at least 1 dose of study drug during the parent study 102 and/or received at least 1 dose of study drug during this Open label study.) | 3 (Cumulative TC Efficacy Set 102/105 included all participants who were randomized to TC ELX/TEZ/IVA and received at least 1 dose of study drug during the parent study 102 and/or received at least 1 dose of study drug during this Open label study. Three participants from parent study 102 (not enrolled in this study) were included in this analysis set.)
Cumulative TC Efficacy Set 103/105 | 107 (Cumulative TC Efficacy Set 103/105 included all participants who were randomized to TC ELX/TEZ/IVA and received at least 1 dose of study drug during the parent study 103 and/or received at least 1 dose of study drug during this Open label study.) | 0
Completed | 354 | 0
Not Completed | 153 | 3
Not completed — Adverse Event | 15 | 0
Not completed — Withdrawal of consent (not due to AE) | 18 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Commercial drug is Available for participant | 48 | 0
Not completed — Death | 1 | 0
Not completed — Other non-compliance | 2 | 0
Not completed — Physician Decision | 6 | 0
Not completed — Other | 58 | 0
Not completed — Enrolled but never dosed | 1 | 0
Not completed — Not enrolled in 105 study | 0 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug in this open label study were included in the baseline characteristics.
Groups:
- ELX/TEZ/IVA: Treatment Period: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 192 weeks.
  Extension Period: Participants from certain countries participated in extension period and continued to received ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the extension period for 48 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 506
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251
  Male | 255
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 460
  Not collected per local regulations | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 470
  Black or African American | 4
  American Indian or Alaska Native | 1
  Other | 3
  Not collected per local regulations | 25
  Multiple | 3

OUTCOME MEASURES:

1. Primary Outcome: Treatment Period: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to Week 196
Population: The Open-Label Safety Set (OL-SS) included all participants who had received at least 1 dose of study drug in this open label study.
Measure: Count of Participants; unit: Participants
Groups:
- ELX/TEZ/IVA: Treatment Period: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 192 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 506
Participants
  Participants With TEAEs | 504
  Participants With SAEs | 175

2. Secondary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 102/105 Efficacy Set
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. This analysis set included study 102 parent study participants who received Placebo-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: OL-FAS is defined as all enrolled participants who received at least 1 dose of study drug in this open label study. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome. Here "Number Analyzed" signifies participants who were evaluable for the specified category. Baseline was defined as the parent study baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Groups:
- ELX/TEZ/IVA: All participants who received Placebo and ELX/TEZ/IVA FDC in parent study 102 were to be administered ELX 200 mg qd/TEZ 100 mg qd /IVA 150 mg q12h in the treatment period for 192 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 269
percentage points
  Placebo-ELX/TEZ/IVA: number analyzed (Participants) | 136
  Placebo-ELX/TEZ/IVA | 15.3 (0.8)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 133
  ELX/TEZ/IVA-ELX/TEZ/IVA | 13.8 (0.8)

3. Secondary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 103/105 Efficacy Set
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. This analysis set included study 103 parent study participants who received TEZ/IVA-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: OL-FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome. Here "Number Analyzed" signifies participants who were evaluable for the specified category. Baseline was defined as the parent study baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Groups:
- ELX/TEZ/IVA: All participants who received TEZ/IVA and ELX/TEZ/IVA FDC in parent study 103 were to be administered ELX 200 mg qd/TEZ 100 mg qd /IVA 150 mg q12h in the treatment period for 192 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 68
percentage points
  TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 32
  TEZ/IVA-ELX/TEZ/IVA | 10.9 (1.3)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 36
  ELX/TEZ/IVA-ELX/TEZ/IVA | 10.7 (1.3)

4. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl) for 102/105 Efficacy Set
Description: Sweat samples were collected using an approved collection device. This analysis set included study 102 parent study participants who received Placebo-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 261
millimole per liter (mmol/L)
  Placebo-ELX/TEZ/IVA: number analyzed (Participants) | 133
  Placebo-ELX/TEZ/IVA | -47.0 (1.6)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 128
  ELX/TEZ/IVA-ELX/TEZ/IVA | -45.3 (1.6)

5. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl) for 103/105 Efficacy Set
Description: Sweat samples were collected using an approved collection device. This analysis set included study 103 parent study participants who received TEZ/IVA-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 69
mmol/L
  TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 31
  TEZ/IVA-ELX/TEZ/IVA | -48.2 (3.8)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 38
  ELX/TEZ/IVA-ELX/TEZ/IVA | -48.2 (3.5)

6. Secondary Outcome: Number of Pulmonary Exacerbations (PEx) for 102/105 Efficacy Set
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: From Baseline at Week 192
Population: Cumulative TC Efficacy Set 102/105 included all participants who were randomized to TC ELX/TEZ/IVA and received at least 1 dose of study drug during the parent study 102 and/or received at least 1 dose of study drug during this open label study. Baseline was defined as the parent study baseline.
Measure: Number; unit: PEx events
Groups:
- ELX/TEZ/IVA: All participants who received Placebo and ELX/TEZ/IVA TC in parent study 102 were to be administered ELX 200 mg qd/TEZ 100 mg qd /IVA 150 mg q12h in the treatment period for 192 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 403
PEx events | 174

7. Secondary Outcome: Number of Pulmonary Exacerbations (PEx) for 103/105 Efficacy Set
Description: as for outcome 6
Time Frame: From Baseline at Week 192
Population: Cumulative TC Efficacy Set 103/105 included all participants who were randomized to TC ELX/TEZ/IVA and received at least 1 dose of study drug during the parent study 103 and/or received at least 1 dose of study drug during this open label study. Baseline was defined as the parent study baseline.
Measure: Number; unit: PEx events
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 107
PEx events | 43

8. Secondary Outcome: Time to First PEx for 102/105 Efficacy Set
Description: Time-to-first pulmonary exacerbation was analyzed using Kaplan-Meier estimates and expressed in terms of event-free probability. PEx was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: From Baseline at Week 192
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 403
days | NA [NA to NA] — Median and 95% confidence interval could not be estimated because less than 50% of participants had events.

9. Secondary Outcome: Time to First PEx for 103/105 Efficacy Set
Description: as for outcome 8
Time Frame: From Baseline at Week 192
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 107
days | NA [NA to NA] — Median and 95% confidence interval could not be estimated because less than 50% of participants had events.

10. Secondary Outcome: Absolute Change in Body Mass Index (BMI) for 102/105 Efficacy Set
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).This analysis set included study 102 parent study participants who received Placebo-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kilogram per meter square (kg/m^2)
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 283
kilogram per meter square (kg/m^2)
  Placebo-ELX/TEZ/IVA: number analyzed (Participants) | 144
  Placebo-ELX/TEZ/IVA | 1.81 (0.16)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 139
  ELX/TEZ/IVA-ELX/TEZ/IVA | 1.74 (0.16)

11. Secondary Outcome: Absolute Change in Body Mass Index (BMI) for 103/105 Efficacy Set
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).This analysis set included study 103 parent study participants who received TEZ/IVA-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 74
kg/m^2
  TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 32
  TEZ/IVA-ELX/TEZ/IVA | 1.72 (0.24)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 42
  ELX/TEZ/IVA-ELX/TEZ/IVA | 1.85 (0.22)

12. Secondary Outcome: Absolute Change in BMI Z-score for 102/105 Efficacy Set
Description: BMI was defined as weight in kg divided by height in m^2. Z-score is a statistical measure to describe whether a mean was above or below the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age z-score. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher BMI. This analysis set included study 102 parent study participants who received Placebo-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: OL-FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were <=20 years of age at Baseline. Here "Number Analyzed" signifies participants who were evaluable for the specified category. Baseline was defined as the parent study baseline.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 57
z-score
  Placebo-ELX/TEZ/IVA: number analyzed (Participants) | 34
  Placebo-ELX/TEZ/IVA | 0.24 (0.09)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 23
  ELX/TEZ/IVA-ELX/TEZ/IVA | 0.18 (0.09)

13. Secondary Outcome: Absolute Change in BMI Z-score for 103/105 Efficacy Set
Description: BMI was defined as weight in kg divided by height in m^2. Z-score is a statistical measure to describe whether a mean was above or below the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age z-score. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher BMI. This analysis set included study 103 parent study participants who received TEZ/IVA-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 15
z-score
  TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 8
  TEZ/IVA-ELX/TEZ/IVA | 0.36 (0.14)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 7
  ELX/TEZ/IVA-ELX/TEZ/IVA | 0.24 (0.15)

14. Secondary Outcome: Absolute Change in Body Weight for 102/105 Efficacy Set
Description: This analysis set included study 102 parent study participants who received Placebo-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 283
kg
  Placebo-ELX/TEZ/IVA: number analyzed (Participants) | 144
  Placebo-ELX/TEZ/IVA | 6.6 (0.5)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 139
  ELX/TEZ/IVA-ELX/TEZ/IVA | 6.0 (0.5)

15. Secondary Outcome: Absolute Change in Body Weight for 103/105 Efficacy Set
Description: This analysis set included study 103 parent study participants who received TEZ/IVA and ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 74
kg
  TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 32
  TEZ/IVA-ELX/TEZ/IVA | 6.1 (0.8)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 42
  ELX/TEZ/IVA-ELX/TEZ/IVA | 6.3 (0.7)

16. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score for 102/105 Efficacy Set
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. This analysis set included study 102 parent study participants who received Placebo-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 295
units on a scale
  Placebo-ELX/TEZ/IVA: number analyzed (Participants) | 148
  Placebo-ELX/TEZ/IVA | 15.3 (1.5)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 147
  ELX/TEZ/IVA-ELX/TEZ/IVA | 18.3 (1.5)

17. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score for 103/105 Efficacy Set
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. This analysis set included study 103 parent study participants who received TEZ/IVA and ELX/TEZ/IVA.
Time Frame: From Baseline at Week 192
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 75
units on a scale
  TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 33
  TEZ/IVA-ELX/TEZ/IVA | 14.8 (2.6)
  ELX/TEZ/IVA-ELX/TEZ/IVA: number analyzed (Participants) | 42
  ELX/TEZ/IVA-ELX/TEZ/IVA | 17.6 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) are reported separately for both Periods. Treatment period covers 1st dose till 196 weeks in treatment period; extension period covers 1st dose in extension period till safety follow-up or end of study, whichever occurs first. The actual total duration for AE collection is up to 222 weeks.
Description: The study was conducted as a treatment period in countries including United States (US) with commercially-available ELX/TEZ/IVA. The regional protocol for other countries without commercially-available ELX/TEZ/IVA was amended so that participants in these countries had the opportunity to participate for up to an additional 48 weeks in extension period. The adverse events data has been reported for both the parts separately.
Groups:
- Treatment Period: ELX/TEZ/IVA: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 192 weeks.
- Extension Period: ELX/TEZ/IVA: Participants from certain countries participated in extension period and continued to receive ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the extension period for 48 weeks.
Arm/Group | Treatment Period: ELX/TEZ/IVA | Extension Period: ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 1/506 | 0/11
Serious Adverse Events (participants affected / at risk) | 175/506 | 0/11
Other Adverse Events (participants affected / at risk) | 501/506 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: ELX/TEZ/IVA (N=506) | Extension Period: ELX/TEZ/IVA (N=11)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 1 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 | 0
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 6 | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 9 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric fistula (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Physical deconditioning (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 1 | 0
Chest wall abscess (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 83 | 0
Influenza (Infections and infestations) | 7 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 3 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fracture of penis (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 0
Bacterial test positive (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Enterovirus test positive (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Human rhinovirus test positive (Investigations) | 1 | 0
Influenza A virus test positive (Investigations) | 2 | 0
Pulmonary function test decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Philadelphia positive acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Miller Fisher syndrome (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Anger (Psychiatric disorders) | 1 | 0
Anorexia nervosa (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 3 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 5 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Testicular torsion (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: ELX/TEZ/IVA (N=506) | Extension Period: ELX/TEZ/IVA (N=11)
Palpitations (Cardiac disorders) | 11 | 1
Abdominal distension (Gastrointestinal disorders) | 31 | 0
Abdominal pain (Gastrointestinal disorders) | 76 | 0
Abdominal pain upper (Gastrointestinal disorders) | 49 | 0
Constipation (Gastrointestinal disorders) | 72 | 0
Diarrhoea (Gastrointestinal disorders) | 89 | 0
Nausea (Gastrointestinal disorders) | 91 | 0
Vomiting (Gastrointestinal disorders) | 67 | 0
Fatigue (General disorders) | 118 | 0
Influenza like illness (General disorders) | 33 | 0
Malaise (General disorders) | 26 | 0
Pain (General disorders) | 37 | 0
Pyrexia (General disorders) | 147 | 0
Immunisation reaction (Immune system disorders) | 83 | 0
Seasonal allergy (Immune system disorders) | 45 | 0
COVID-19 (Infections and infestations) | 168 | 0
Cystitis (Infections and infestations) | 8 | 1
Gastroenteritis (Infections and infestations) | 31 | 0
Hordeolum (Infections and infestations) | 18 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 224 | 3
Influenza (Infections and infestations) | 63 | 0
Lower respiratory tract infection (Infections and infestations) | 7 | 1
Nasopharyngitis (Infections and infestations) | 154 | 0
Pharyngitis (Infections and infestations) | 37 | 0
Rhinitis (Infections and infestations) | 50 | 0
Sinusitis (Infections and infestations) | 76 | 1
Upper respiratory tract infection (Infections and infestations) | 120 | 1
Urinary tract infection (Infections and infestations) | 43 | 0
Viral upper respiratory tract infection (Infections and infestations) | 36 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 27 | 0
Procedural pain (Injury, poisoning and procedural complications) | 21 | 1
Alanine aminotransferase increased (Investigations) | 72 | 0
Aspartate aminotransferase increased (Investigations) | 68 | 0
Bacterial test positive (Investigations) | 50 | 0
Blood bilirubin increased (Investigations) | 31 | 0
Blood creatine phosphokinase increased (Investigations) | 72 | 0
Gamma-glutamyltransferase increased (Investigations) | 26 | 0
Pulmonary function test decreased (Investigations) | 30 | 0
SARS-CoV-2 test positive (Investigations) | 45 | 0
Weight decreased (Investigations) | 32 | 0
Decreased appetite (Metabolism and nutrition disorders) | 26 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 33 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 71 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 51 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 33 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 0
Dizziness (Nervous system disorders) | 38 | 0
Headache (Nervous system disorders) | 178 | 0
Anxiety (Psychiatric disorders) | 38 | 0
Depression (Psychiatric disorders) | 40 | 0
Insomnia (Psychiatric disorders) | 34 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 231 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 82 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 37 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 113 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 166 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 61 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 33 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 76 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 62 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 127 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 33 | 0
Acne (Skin and subcutaneous tissue disorders) | 49 | 0
Rash (Skin and subcutaneous tissue disorders) | 57 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT03525574/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT03525574/SAP_001.pdf